CLINICAL TRIAL: NCT07107698
Title: Accuracy of Non-Invasive Blood Pressure Monitoring During Video-Assisted Thoracoscopic Surgery With One-Lung Ventilation: A Prospective Error Grid Analysis
Brief Title: Blood Pressure Monitoring Accuracy in Patients Undergoing Lung Surgery With One-Lung Ventilation Using an Arm Cuff and Arterial Line
Status: Not yet recruiting | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Principal Investigator, Kamil Darcin, Associate professor, Koç University
Other Study IDs: 2025.244.IRB2.110
Record Dates: First submitted 2025-07-30; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Non-Invasive Blood Pressure Monitoring During Thoracoscopic Surgery With One-Lung Ventilation
Keywords: Non-invasive blood pressure; Invasive arterial pressure; Thoracoscopic surgery; One-lung ventilation; Intraoperative monitoring; Error grid analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Surgical Cohort: Adults (18 years and older) undergoing video-assisted thoracoscopic surgery (VATS) with one-lung ventilation who are already scheduled to receive invasive arterial blood pressure monitoring as part of routine clinical care. Participants will have paired invasive and non-invasive blood pressure measurements recorded during surgery for comparison using error grid analysis.

SUMMARY:
This study will test how accurate a blood pressure cuff is during a specific type of chest surgery.

In some lung surgeries, doctors use a method called video-assisted thoracoscopic surgery (VATS), where small tools and a camera are inserted through the chest wall. During these procedures, patients often have only one lung ventilated to give the surgeon more space to work. This setup can affect how well a blood pressure cuff on the arm reflects the true blood pressure inside the body.

This study will compare readings from the arm cuff (non-invasive) with those from a thin tube placed inside an artery (invasive), which is more accurate but also more uncomfortable and carries some risks.

Researchers will use a method called error grid analysis to see how closely the cuff readings match the invasive ones. They want to find out if the cuff is accurate enough to be used safely in these surgeries. If it is, patients might not need an invasive line as often in the future.

People 18 years or older who are already going to have invasive blood pressure monitoring during planned thoracic surgery with one-lung ventilation may be able to join the study. The research team will collect blood pressure measurements about every 20 minutes during surgery, as well as basic information like age, weight, and what medications are given.

DETAILED DESCRIPTION:
This is a prospective observational study designed to evaluate the clinical accuracy and reliability of non-invasive blood pressure (NIBP) monitoring in adult patients undergoing video-assisted thoracoscopic surgery (VATS) with one-lung ventilation (OLV). The accuracy of NIBP will be assessed by comparing it to invasive arterial blood pressure (IABP), which is considered the reference standard. The comparison will be performed using error grid analysis, a method that not only quantifies measurement differences but also categorizes the clinical risk of those discrepancies.

During VATS procedures, one lung is intentionally deflated to improve surgical access, which alters thoracic pressures, ventilation dynamics, and cardiovascular physiology. These changes may affect the accuracy of peripheral blood pressure measurements obtained using an arm cuff. Previous evaluations of NIBP in surgical patients have primarily relied on Bland-Altman analysis, which measures statistical agreement but does not assess the clinical consequences of disagreement between methods.

Error grid analysis overcomes this limitation by mapping paired NIBP and IABP values into predefined clinical risk zones (A-E), based on their potential to affect treatment decisions. Zone A represents measurements with no risk of causing inappropriate treatment, while Zones B through E indicate increasing levels of clinical risk due to measurement error.

In this study, NIBP and IABP measurements will be recorded simultaneously approximately every 20 minutes throughout surgery. The percentage of measurements that fall within each error grid zone will be calculated. If fewer than 90% of the paired measurements fall within Zone A, NIBP will be considered insufficiently reliable for use without concurrent invasive monitoring in this clinical context.

A pilot study of five patients was used to estimate the intracluster correlation coefficient and design effect, which informed the final sample size calculation. Based on these preliminary data, a total sample size of 90 patients is estimated to provide adequate statistical power to evaluate the primary outcome with 95% confidence and a 5% margin of error.

The study will also collect intraoperative data that may influence blood pressure measurement accuracy, such as the use of vasoactive infusions. These data may help identify subgroups in which NIBP is more or less reliable during one-lung ventilation.

The results of this study may help refine intraoperative monitoring strategies and potentially reduce unnecessary use of invasive blood pressure lines in selected thoracic surgical patients, improving both safety and comfort while maintaining clinical reliability.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Scheduled to undergo video-assisted thoracoscopic surgery with one-lung ventilation
* Will receive invasive arterial blood pressure monitoring as part of routine clinical care

Exclusion Criteria:

* Has peripheral artery disease
* Has congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be selected from adult patients scheduled for video-assisted thoracoscopic surgery with one-lung ventilation at Koç University Hospital, a tertiary care academic medical center in Istanbul, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of Paired Systolic Blood Pressure Measurements Within Zone A of the Error Grid | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of systolic non-invasive blood pressure (NIBP) measurements that fall within Zone A of the consensus error grid with calibrated risk zones, as described by Saugel et al.[1]. Zone A represents measurement pairs with no risk of leading to inappropriate clinical decisions, based on comparison with simultaneously recorded systolic invasive arterial blood pressure values. Systolic NIBP measurements will be considered acuurate if 90% or more of the paired values fall within Zone A.
  1. Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185
Proportion of Paired Mean Arterial Pressure (MAP) Measurements Within Zone A of the Error Grid | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of non-invasive mean arterial pressure (MAP) measurements that fall within Zone A of the consensus error grid with calibrated risk zones, as described by Saugel et al.[1]. Zone A represents measurement pairs with no risk of leading to inappropriate clinical decisions, based on comparison with simultaneously recorded invasive MAP values. Non-invasive MAP measurements will be considered accurate if 90% or more of the paired values fall within Zone A.
  1. Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185

SECONDARY OUTCOMES:
Distribution of Paired Systolic Blood Pressure Measurements Across All Error Grid Zones (A-E) | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of paired systolic blood pressure measurements that fall into each zone (A, B, C, D, E) of the consensus error grid. Error grid zones reflect the clinical risk of acting on the non-invasive measurement: Zone A: No risk Zone B: Low risk Zone C: Moderate risk Zone D: Significant risk of undertreatment Zone E: Significant risk of overtreatment The distribution will be reported as the percentage of all paired measurements falling into each zone.
Distribution of Paired Mean Arterial Pressure (MAP) Measurements Across All Error Grid Zones (A-E) | Intraoperative period (measurements taken every 20 minutes during surgery)
  The percentage of paired mean arterial pressure (MAP) measurements that fall into each zone (A through E) of the consensus error grid. Error grid zones reflect the clinical risk of acting on the non-invasive measurement: Zone A: No risk Zone B: Low risk Zone C: Moderate risk Zone D: Significant risk of undertreatment Zone E: Significant risk of overtreatment The distribution will be reported as the percentage of all paired measurements falling into each zone.
Effect of Antihypertensive Medication Use on the Accuracy of Systolic NIBP Measurements | Intraoperative period (measurements taken every 20 minutes during surgery)
  This outcome compares the likelihood that individual systolic non-invasive blood pressure (NIBP) measurements fall within Zone A of the consensus error grid between participants who use antihypertensive medications and those who do not. Zone A indicates values that would not lead to inappropriate clinical decisions. To account for the fact that multiple blood pressure measurements are collected from each participant, the analysis will use mixed-effects logistic regression. This model includes a random effect for each participant to account for the correlation among repeated measurements within the same individual.
Effect of Antihypertensive Medication Use on the Accuracy of Mean Arterial Pressure (MAP) NIBP Measurements | Intraoperative period (measurements taken every 20 minutes during surgery)
  This outcome compares the likelihood that individual non-invasive mean arterial pressure (MAP) measurements fall within Zone A of the consensus error grid between participants with and without antihypertensive medication use. Zone A represents measurement pairs that are clinically acceptable. To account for the fact that multiple blood pressure measurements are collected from each participant, the analysis will use mixed-effects logistic regression. This model includes a random effect for each participant to account for the correlation among repeated measurements within the same individual.

CONTACTS AND LOCATIONS:
Overall Officials: Kamil Darcin, Associate professor, Study Director — Koç University School of Medicine

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual participant data (IPD) that underlie the results of the study will be shared. These data will be made publicly available through the Zenodo repository following study completion and publication.
Supporting Information: Study Protocol
Time Frame: Beginning at the time of the first publication of study results, with no end date.
Access Criteria: The anonymized individual participant data (IPD) and supporting documentation will be openly available to the public via the Zenodo data repository. No proposal, request, or data use agreement is required. Researchers may download the dataset directly from Zenodo upon publication. The data are intended for secondary analysis, validation of findings, or meta-research. A citation to the original study publication and dataset DOI is requested when using the data.
URL: https://zenodo.org/

REFERENCES:
- [Background] Saugel B, Grothe O, Nicklas JY. Error Grid Analysis for Arterial Pressure Method Comparison Studies. Anesth Analg. 2018 Apr;126(4):1177-1185. doi: 10.1213/ANE.0000000000002585. PMID 29239945